CLINICAL TRIAL: NCT04880499
Title: Emacrit Plus in Prosthetic Hip and Knee Surgery
Brief Title: Iron and Vitamin Supplementation in Hip/Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EMA-IRON (PI: M Briguglio); L4143 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Orthopedic Disorder; Hip Arthropathy; Knee Arthropathy; Anemia; Iron Poor Blood
MeSH Terms: conditions — Musculoskeletal Diseases; Anemia | interventions — Iron; Folic Acid; Riboflavin; Vitamin B 12

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (group A) (Experimental): Patients who are subjected to the intervention, being iron plus other cofactors for hematopoiesis, other than the standard of care.
  Interventions: Dietary Supplement: Iron plus folic acid, vitamin B2, B6, B12, C, and E
- Control (group B) (No Intervention): Patients who are not subjected to the intervention and follow the standard of care.

INTERVENTIONS:
Dietary Supplement: Iron plus folic acid, vitamin B2, B6, B12, C, and E — A number of 30 subjects are supplemented with iron plus folic acid, vitamin B2, B6, B12, C, and E daily for 60+/-15 days before orthopedic surgery.
  Arms: Intervention (group A)

SUMMARY:
Randomized controlled trial to evaluate the efficacy of oral iron supplementation plus cofactors in reducing the prevalence of preoperative anemia in a cohort of 60 patients undergoing elective prosthetic hip or knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* ASA 1, 2, or 3
* No neuropsychiatric conditions
* Acceptance of informed consent
* Elective prosthetic hip or knee surgery

Exclusion Criteria:

* ASA 4
* Present or past neuropsychiatric conditions
* Hip or knee revision surgery
* Use of iron as dietary supplement
* Known erythrocytosis
* Incompatible hypersensitivities
* Iron metabolism disorders
* Lymphoproliferative disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Change of blood hemoglobin levels | Baseline and 60 days +/- 15 days
  Change of hemoglobin concentration (g/dl) from baseline and after 60 days +/- 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Briguglio, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided